CLINICAL TRIAL: NCT03913221
Title: Pharmacokinetics and Safety of Caffeine in Neonates With Hypoxic-Ischemic Encephalopathy
Brief Title: Caffeine for Hypoxic-Ischemic Encephalopathy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 19-0348
Record Dates: First submitted 2019-04-10; First posted 2019-04-12 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-01

CONDITIONS: Hypoxic-Ischemic Encephalopathy
MeSH Terms: conditions — Hypoxia-Ischemia, Brain | interventions — caffeine citrate

STUDY DESIGN:
Intervention Model Description: The first cohort of 9 infants will receive a lower maintenance dose of caffeine. Following a safety review, an additional 9 infants will receive a higher maintenance dose.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Low Dose Caffeine (5 mg/kg) (Active Comparator): Within 24 hours of delivery, participants will receive low dose administration of Caffeine citrate.
  Interventions: Drug: Caffeine Citrate 5 mg/kg
- High Dose Caffeine (10 mg/kg) (Active Comparator): Within 24 hours of delivery, participants will receive high dose administration of Caffeine citrate.
  Interventions: Drug: Caffeine Citrate 10 mg/kg

INTERVENTIONS:
Drug: Caffeine Citrate 5 mg/kg — Loading dose of caffeine 20 mg/kg IV followed by two daily doses of 5 mg/kg IV.
  Other Names: Cafcit
  Arms: Low Dose Caffeine (5 mg/kg)
Drug: Caffeine Citrate 10 mg/kg — Loading dose of caffeine 20 mg/kg IV followed by two daily doses of 10 mg/kg IV.
  Other Names: Cafcit
  Arms: High Dose Caffeine (10 mg/kg)

SUMMARY:
Hypoxic-ischemic encephalopathy (HIE) due to perinatal asphyxia is common and often fatal. Therapeutic hypothermia reduces mortality and morbidity in infants with HIE. Even with the widespread use of therapeutic hypothermia, ~60% of infants with HIE die or have neurodevelopmental impairment. As a result, there is an urgent, unmet public health need to develop adjuvant therapies to improve survival and neurodevelopmental outcomes in this population.

Caffeine may offer neuroprotection for infants with HIE by blocking adenosine receptors in the brain and reducing neuronal cell death. In animal models of HIE, caffeine reduces white matter brain injury. Drugs in the same class as caffeine (i.e., methylxanthines) have been shown to be protective against acute kidney injury in the setting of HIE. However, their safety and efficacy have not been studied in the setting of therapeutic hypothermia and their effect on neurological outcomes is not known. Since these drugs reduce injury to the kidney in infants with HIE, they may also reduce injury to the brain.

This phase I study will evaluate the pharmacokinetics, safety, and preliminary effectiveness of caffeine as an adjuvant therapy to improve neurodevelopmental outcomes in infants with HIE.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent from parent or guardian
* ≥ 36 weeks gestational age at birth
* Receiving therapeutic hypothermia for a diagnosis of HIE
* Intravenous (IV) access
* Postnatal age < 24 hours

Exclusion Criteria:

* Receiving > 1 anti-epileptic drug for seizures
* Sustained (>4 hours) heart rate > 180 beats per minute
* Known major congenital anomaly
* Any condition which would make the participant, in the opinion of the investigator, unsuitable for the study

Max Age: 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2019-08-14 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wesley M Jackson, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- The University of North Carolina at Chapel Hill Newborn Critical Care Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata.

REFERENCES:
- [Background] Shankaran S, McDonald SA, Laptook AR, Hintz SR, Barnes PD, Das A, Pappas A, Higgins RD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Neonatal Magnetic Resonance Imaging Pattern of Brain Injury as a Biomarker of Childhood Outcomes following a Trial of Hypothermia for Neonatal Hypoxic-Ischemic Encephalopathy. J Pediatr. 2015 Nov;167(5):987-93.e3. doi: 10.1016/j.jpeds.2015.08.013. Epub 2015 Sep 16. PMID 26387012
- [Background] Shankaran S, Laptook AR, Ehrenkranz RA, Tyson JE, McDonald SA, Donovan EF, Fanaroff AA, Poole WK, Wright LL, Higgins RD, Finer NN, Carlo WA, Duara S, Oh W, Cotten CM, Stevenson DK, Stoll BJ, Lemons JA, Guillet R, Jobe AH; National Institute of Child Health and Human Development Neonatal Research Network. Whole-body hypothermia for neonates with hypoxic-ischemic encephalopathy. N Engl J Med. 2005 Oct 13;353(15):1574-84. doi: 10.1056/NEJMcps050929. PMID 16221780
- [Result] Jackson W, Gonzalez D, Greenberg RG, Lee YZ, Laughon MM. A phase I trial of caffeine to evaluate safety in infants with hypoxic-ischemic encephalopathy. J Perinatol. 2024 Apr;44(4):508-512. doi: 10.1038/s41372-023-01752-y. Epub 2023 Aug 16. PMID 37587184

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 17 infants undergoing therapeutic hypothermia for hypoxic ischemic encephalopathy were enrolled at the University of North Carolina at Chapel Hill Newborn Critical Care Center between August 2019 and December 2022.
Period: Low Dose Cohort
Arm/Group | Low Dose Caffeine (5 mg/kg) | High Dose Caffeine (10 mg/kg)
Started | 9 | 0
Completed | 9 | 0
Not Completed | 0 | 0
Period: High Dose Cohort
Arm/Group | Low Dose Caffeine (5 mg/kg) | High Dose Caffeine (10 mg/kg)
Started | 0 | 8
Completed | 0 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose Caffeine (5 mg/kg) | High Dose Caffeine (10 mg/kg) | Total
Number analyzed (Participants) | 9 | 8 | 17
Age, Customized [Count of Participants; unit: Participants]
  >/= 36 weeks gestational age | 9 | 8 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 9 | 5 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 3 | 8
  White | 3 | 5 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: Area Under Plasma Concentration-time at Time t (AUC0-t) for Caffeine
Description: AUC0-t defines area under the plasma concentration-time curve (AUC) from administration to the last quantifiable concentration at time t.
Time Frame: 7 samples will be collected with the following optimal sampling windows: 0-15 minutes, 30-60 minutes, 1-3 hours, 3-6 hours, 6-12 hours, 12-18 hours, 15 minutes prior to next dose.
Measure: Mean (Standard Deviation); unit: mg*hr/L
Arm/Group | Low Dose Caffeine (5 mg/kg) | High Dose Caffeine (10 mg/kg)
Number analyzed (Participants) | 9 | 8
mg*hr/L
  AUC (0-72) | 1137.36 (324.96) | 1177.94 (134.42)
  AUC (0-infinity) | 2213.26 (540.81) | 2768.25 (338.06)

2. Secondary Outcome: Number of Participants With Seizures Requiring >1 Anti-Epileptic Medication
Description: As a potential complication of caffeine exposure, seizure activity requiring >1 anti-epileptic medication is reported.
Time Frame: From the first dose of caffeine to 7 days following the final dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Caffeine (5 mg/kg) | High Dose Caffeine (10 mg/kg)
Number analyzed (Participants) | 9 | 8
Participants | 1 | 0

3. Secondary Outcome: Number of Participants With Necrotizing Enterocolitis
Description: As a potential complication of caffeine exposure, the number of participants with necrotizing enterocolitis defined as Bell Stage II or III are reported.
Time Frame: From the first dose of caffeine to 7 days following the final dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Caffeine (5 mg/kg) | High Dose Caffeine (10 mg/kg)
Number analyzed (Participants) | 9 | 8
Participants | 0 | 0

4. Secondary Outcome: Number of Participants With Abnormal MRI Brain Findings Based on NICHD Neonatal Research Network Score
Description: The National Institute of Child Health and Human Development (NICHD) Neonatal Research Network developed and validated an MRI scoring system that categorizes severity of brain injury in the Trial of Hypothermia for Neonatal Hypoxic-Ischemic Encephalopathy. A higher score is considered a worse outcome.
  * Score 0: Normal T2 MRI
  * Score 1A: Minimal cerebral lesions only with involvement of basal ganglia, thalamus
  * Score 1B: Extensive cerebral lesions
  * Score 2A: Basal ganglia thalamic, anterior or posterior limb of internal capsule, or watershed infarction
  * Score 2B: 2A with cerebral lesions
  * Score 3: Hemispheric devastation
Time Frame: During initial hospitalization, approximately 7-14 postnatal days
Population: Two infants died during hospitalization and did not have MRI performed.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Caffeine (5 mg/kg) | High Dose Caffeine (10 mg/kg)
Number analyzed (Participants) | 8 | 7
Participants
  Score 0 | 3 | 2
  Score 1A | 2 | 2
  Score 1B | 1 | 3
  Score 2A | 0 | 0
  Score 2B | 2 | 0
  Score 3 | 0 | 0

5. Secondary Outcome: Number of Participants With a Bayley Scales of Infant Development (BSID-III) Cognitive, Language, or Motor Composite Score < 85
Description: The BSID-III is a series of measurements to assess the motor (fine and gross), language (receptive and expressive), and cognitive development of infants and toddlers and consists of a series of developmental play tasks. The composite scores are scaled to a metric with a range of 40 to 160, a mean of 100, and a standard deviation of 15. Therefore, children with a composite score < 85 are 1 standard deviation below the mean in that area.
Time Frame: 18-24 months of age
Population: Bayley-III examinations were planned at the beginning of the study per institutional standard of care. However, during the study period, clinical practice changed, and due to COVID-19 pandemic-related staff turnover, Bayley-III examinations were no longer routinely obtained in Hypoxic-ischemic encephalopathy (HIE) patients. As Bayley-III exams were not included in the study budget and were not a primary study aim, these data were not collected. The protocol was not amended with this change.
Arm/Group | Low Dose Caffeine (5 mg/kg) | High Dose Caffeine (10 mg/kg)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From the first dose of study intervention through 7 days after the last dose of study intervention, approximately 10 days.
Arm/Group | Low Dose Caffeine (5 mg/kg) | High Dose Caffeine (10 mg/kg)
All-Cause Mortality (participants affected / at risk) | 1/9 | 1/8
Serious Adverse Events (participants affected / at risk) | 3/9 | 2/8
Other Adverse Events (participants affected / at risk) | 8/9 | 4/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose Caffeine (5 mg/kg) (N=9) | High Dose Caffeine (10 mg/kg) (N=8)
Extracorporeal membrane oxygenation (ECMO) (Surgical and medical procedures) | 2 (2) | 1 (1)
Seizures (Nervous system disorders) | 1 (1) | 0 (0) — Seizures requiring more than 1 anti-convulsant medication
Bowel perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose Caffeine (5 mg/kg) (N=9) | High Dose Caffeine (10 mg/kg) (N=8)
Acute Kidney Injury (Renal and urinary disorders) | 2 (2) | 1 (1)
Hepatic Dysfunction (Hepatobiliary disorders) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (5) | 2 (2)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Supraventricular Tachycardia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Subcutaneous Fat Necrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Disseminated Intrvascular Coagulopathy (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Direct Hyperbilirubinemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Seizures (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-26): https://cdn.clinicaltrials.gov/large-docs/21/NCT03913221/Prot_SAP_000.pdf